CLINICAL TRIAL: NCT03893643
Title: Multicentre Prospective Observational Study: Resentment of Mucocutaneous Manifestations and the Value of Dermatological Examination in the Early Detection of Type 2 Neurofibromatosis in Children Under 15 Years of Age
Brief Title: Cutaneous and Mucosal Manifestations of Neurofribromatosis Type 2 in Children Under 15
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 18-DERMATO-01
Record Dates: First submitted 2019-01-21; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-01

CONDITIONS: Neurofibromatosis 2; Dermatology/Skin - Other
MeSH Terms: conditions — Neurofibromatosis 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric population: Pediatric population aged 0 to 15 years with neurofibromatosis type 2
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention in an observational study

SUMMARY:
.Neurofibromatosis type 2 is an inherently autosomal dominant genetic disease, but cases of mosaicism or de novo mutation are not uncommon. the prevalence is estimated at 1 / 60,000. the clinical presentation is based on the appearance of tumors in the central and peripheral nervous system. The current average age of diagnosis is around 25 to 30 years depending on the studies. Currently, the diagnostic criteria are based on the ENT, neurological and opthalmological manifestations of the disease. Cutaneous manifestations have been described in these patients. Except now, mucocutaneous manifestations of the disease are not taken into account for depisatage or diagnosis.

The purpose of this study would be to identify the different cutaneous and mucosal manifestations in a pediatric population under 15 years of age, and to analyze whether this might be of interest in early detection of the disease in association with other symptoms.

ELIGIBILITY:
Inclusion Criteria:

* age up to 15 years
* diagnosis of neurofibromatosis type 2

Exclusion Criteria:

* refusal to participate in the study
* informed consent that can not be obtained because of a disability or difficulties with a - language barrier

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with neurofibromatosis type 2
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
number of cutaneo-mucous lesions present in children with neurofibromatosis type 2 | 3 years
  number of cutaneo-mucous lesions obtain after complete dermatological clinical examination ; if possible take photographs for publication with the patient's consent ; histological results if cutaneous biopsies were performed outside the study

SECONDARY OUTCOMES:
number and type of neurological manifestations. | 3 years
  number and type of neurological clinical data, clinical examination
number and type of descriptioin of ENT manifestations. | 3 years
  number and type of ENT clinical data, clinical examination
number and type of ophthalmological manifestations. | 3 years
  number and type of ophtalmologic clinical data, clinical examination

CONTACTS AND LOCATIONS:
Locations (1):
- Nice Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No